CLINICAL TRIAL: NCT05600491
Title: A Phase III Study of Postoperative Early Temozolomide Treatment Plus STUPP Regimen for Newly Diagnosed GBM Multiforme
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonggao Mou, Professor and Chair, Department of Neurosurgery, Sun Yat-sen University, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Yonggao Mou
Record Dates: First submitted 2022-10-27; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Anaplastic Oligoastrocytoma; Glioblastoma
Keywords: Glioblastoma Multiforme; chemotherapy; Temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Early TMZ chemotherapy (Experimental): Patients were treated with standard concomitant radiochemotherapy regimen (Stupp) plus early postsurgical temozolomide.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Two weeks after surgery, temozolomide was administered orally at 200 mg·m-2 ·d -1 for 5 days. From day 29, patients were treated with a standard therapy regimen (Stupp).
  Other Names: Temodar; TMZ

SUMMARY:
This study was to explore the effectiveness and safety of early TMZ chemotherapy between surgery and chemoradiotherapy plus the standard concomitant radiochemotherapy regimen.

DETAILED DESCRIPTION:
This study was to explore the effectiveness and safety of early temozolomide chemotherapy between surgery and chemoradiotherapy plus the standard concomitant radiochemotherapy regimen. Patients were treated with a standard therapy regimen (Stupp) plus early postsurgical temozolomide.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 years to 70 years; Newly diagnosed Glioblastoma in the supratentorial cerebral hemisphere; Gross total resection or large resection of >70% in imaging studies; Eastern Cooperative Oncology Group performance status of 0-2; Adequate bone marrow, liver and renal function; Ability of subject to understand character and individual consequences of the clinical trial Written informed consent; anticipating survival ≥7 months.

Exclusion Criteria:

Refusal to participate the study; Current diagnosis or history of malignancies within the 3-year period preceding enrollment; Recurrent or multiple malignant gliomas, including gliomatosis cerebri, or metastatic extracalvarial or subtentorial lesions; Known hypersensitivity or contraindication to temozolomide; Pregnant or lactating females; Malignant tumor other than brain tumor; Contraindicated for MRI examination; Unable to comply with the follow-up studies of this trial; Uncontrolled psychotic disorders or epilepsy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-11-08 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5-year
  Overall survival

SECONDARY OUTCOMES:
Progression free survival | 5-year
  Progression free survival
Time to Deterioration (TTD) in Global Health Status/Health Related Quality of Life According to European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) v3.0 in All Randomized Participants | 5-year
  Time to Deterioration (TTD) in Global Health Status/Health Related Quality of Life According to European Organisation for Research and Treatment of Cancer (EORTC) Quality-of-Life Questionnaire Core 30 (QLQ-C30) v3.0 in All Randomized Participants

CONTACTS AND LOCATIONS:
Overall Officials: Mou Y Gao, MD, PhD, Principal Investigator — Department of Neurosurgery/Neuro-oncology, Sun Yat-sen University Cancer Center
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China